CLINICAL TRIAL: NCT06016972
Title: A Randomized, Multi-site, Double-masked Study Evaluating the Safety and Tolerability of QLS-111 Vs Vehicle in Primary Open-angle Glaucoma or Ocular Hypertension Patients
Brief Title: Qlaris Phase 2 Study of QLS-111 in POAG And/or OHT Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QC-111-201; Osprey (Other: Qlaris Bio, Inc.)
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Primary Open Angle Glaucoma (POAG); Primary Open Angle Glaucoma of Both Eyes; Primary Open-Angle Glaucoma, Unspecified Eye; Ocular Hypertension (OHT)
Keywords: Qlaris; POAG; OHT; IOP; Glaucoma; Osprey
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Intervention Model Description: Multi site double masked, vehicle-controlled, randomized, prospective parallel study of 7 days' QAM dosing, followed by 7 days' QPM dosing, and 7 days' BID dosing (7 days of dosing per regimen [21-day treatment period])of an investigational product (IP), QLS-111 or vehicle. Both eyes (OU) will be dosed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, Investigators and their staff, and Sponsor personnel involved with the conduct and monitoring of the study will be masked to the IP identity until after the final database is locked. IP will be provided in identical packaging. Unmasked statistician preparing the masked randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLS-111 ophthalmic solution (Experimental): Qlaris' investigational product, QLS-111 ophthalmic solution, provided in 3 concentrations for this study (0.015%, 0.03%. and 0.075%), single use vials, masked, and preservative free (PF).
  Interventions: Drug: Experimental: QLS-111 ophthalmic solution, (0.015%); Drug: Experimental: QLS-111 ophthalmic solution, (0.03%); Drug: Experimental: QLS-111 ophthalmic solution, (0.075%)
- QLS-111 ophthalmic vehicle solution (Placebo Comparator): Inactive control (0.00%). QLS-111 ophthalmic vehicle solution, single use vials, masked, PF.
  Interventions: Other: QLS-111 ophthalmic vehicle solution

INTERVENTIONS:
Drug: Experimental: QLS-111 ophthalmic solution, (0.015%) — QLS-111 ophthalmic solution, (0.015%) applied QAM OU for 7 days followed by QPM dosing OU for 7 days, and BID OU dosing for 7 days to constitute a 21-day study treatment period. All IP for this study will be supplied masked in PF single use vials.
  Other Names: QLS-111
  Arms: QLS-111 ophthalmic solution
Drug: Experimental: QLS-111 ophthalmic solution, (0.03%) — QLS-111 ophthalmic solution, (0.03%) applied QAM OU for 7 days followed by QPM dosing OU for 7 days, and BID OU dosing for 7 days to constitute a 21-day study treatment period. All IP for this study will be supplied masked in PF single use vials.
  Other Names: QLS-111
  Arms: QLS-111 ophthalmic solution
Drug: Experimental: QLS-111 ophthalmic solution, (0.075%) — QLS-111 ophthalmic solution, (0.075%) applied QAM OU for 7 days followed by QPM dosing OU for 7 days, and BID OU dosing for 7 days to constitute a 21-day study treatment period. All IP for this study will be supplied masked in PF single use vials.
  Other Names: QLS-111
  Arms: QLS-111 ophthalmic solution
Other: QLS-111 ophthalmic vehicle solution — Vehicle ophthalmic solution applied QAM OU for 7 days followed by QPM dosing OU for 7 days, and BID OU dosing for 7 days to constitute a 21-day study treatment period. All IP for this study will be supplied masked in PF single use vials.
  Other Names: vehicle; placebo
  Arms: QLS-111 ophthalmic vehicle solution

SUMMARY:
Qlaris' Phase 2 clinical trial investigating the safety, tolerability, and ocular hypotensive efficacy of QLS-111 in primary open-angle glaucoma (POAG) or ocular hypertension patients.

DETAILED DESCRIPTION:
A randomized, active- and vehicle-controlled, multi-site, double-masked study to evaluate the safety and tolerability of QLS-111 versus vehicle in subjects with primary open-angle glaucoma or ocular hypertension. Primary objective is to evaluate the ocular and systemic safety and tolerability of 3 concentrations of QLS-111 compared to vehicle control. Secondary objective is to evaluate the ocular hypotensive efficacy of 3 concentrations of QLS-111 with once daily morning (QAM), once daily evening (QPM), and twice daily (BID) dosing versus vehicle with QAM, QPM, and BID dosing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to provide written acknowledgement of giving informed consent
* Best corrected visual acuity (BCVA) 20/200 or better Bilateral POAG or OHT with documented historic IOP value(s) ≥24 mmHg, in either eye
* Post-washout IOP ≥22 mmHg in morning on Visits 2 and 3 and ≥18 mmHg at noon on Visit 2

Exclusion Criteria:

* IOP >34 mmHg
* Severe glaucomatous damage that would preclude safe washout of prescribed ocular hypotensive medications
* Previous glaucoma surgery, certain procedures (trabeculotomy, shunt/tubes, cyclodestructive procedure) (selective laser trabeculoplasty (SLT) allowed if done no earlier than 1 year from study, some minimally invasive glaucoma surgeries are allowed if done no earlier than 1 year from study)
* Ocular trauma, ocular infections, ocular inflammation, herpes simplex keratitis of eye
* Use of other ophthalmic concomitant medications during the study
* Uncontrolled hypertension or hypotension
* Significant systemic or psychiatric disease
* Participation in other investigational trial 30 days prior to screening or previous enrollment and treatment with Qlaris investigational product
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular symptoms and ocular treatment-emergent adverse events (TEAEs) | 21 days
  Ocular safety and tolerability: adverse events (AEs)
Clinically significant change in visual acuity | 21 days
  Ocular safety and tolerability: visual acuity
Clinically significant change in findings on slit lamp exam | 21 days
  Ocular safety and tolerability: slit lamp
Clinically significant change in findings on fundus exam | 21 days
  Ocular safety and tolerability: fundus
Incidence of systemic TEAEs | 21 days
  Systemic safety and tolerability: AEs
Clinically significant changes in blood pressure (BP) | 21 days
  Systemic safety and tolerability: vital signs
Clinically significant changes in heart rate (HR) | 21 days
  Systemic safety and tolerability: vital signs

SECONDARY OUTCOMES:
Change from baseline (CFB) of diurnal intraocular pressure (IOP) in the study eye | 21 days
  Ocular hypotensive efficacy: diurnal IOP CFB
CFB in IOP at various timepoints in the study eye | up to 21 days
  Ocular hypotensive efficacy: CFB for multiple timepoints throughout day

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brandano, Study Director — Qlaris Bio, Inc.
Locations (1):
- Coastal Research Associates, LLC, Roswell, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website, pipeline — https://qlaris.bio